CLINICAL TRIAL: NCT04343820
Title: Delayed Breast Reconstruction by Prepectoral Implant After Lipo-preparation : Feasibility, Complications, Evaluation of Aesthetic Result and Quality of Life.
Brief Title: Delayed Breast Reconstruction by Prepectoral Implant After Lipo-preparation (RM2prepec)
Acronym: RM2prepec
Status: Active, not recruiting | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-N-2018-15
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Female
Keywords: reconstruction; lipo-modelling; breast cancer; mastectomy; prepectoral implant
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast reconstruction: Women who have had a mastectomy and want a secondary breast reconstruction by implant.
  Interventions: Procedure: Breast reconstruction

INTERVENTIONS:
Procedure: Breast reconstruction — Breast reconstruction by prepectoral positioned implant after lipo-preparation of the wall.

SUMMARY:
Breast implants associated with the installation of a complementary matrix (of dermal or synthetic origin), showed satisfactory results in term of post-operative follow-up but also aesthetic outcomes.

The objective of the subcutaneous positioning of this implant, is to reduce the muscular pain related to the stretching of the muscular muscle, the deformations related to the muscular contraction with an animation of the prothesis, but also the risk of hull when associated with a matrix. It also pursues the objective, of obtaining a better aesthetic result, by systematically coupling at least one lipo-modelling session.

For a long time, patients with a history of mastectomy and radiotherapy benefited from secondary breast flap reconstruction, in order to reduce the risk of complications and achieve a satisfying aesthetic outcome. But the lipo-filling technique allowed to reconsider the management of these patients.

The benefits of fat tissue transplants are know to improve tissue trophicity (flexibility, thickness, vascularization).

The objective of this study, is to evaluate the feasibility of secondary breast reconstructions by prepectoral positioned implant after lipo-preparation of the wall.

DETAILED DESCRIPTION:
60 women who have had a mastectomy and want a secondary breast reconstruction by implant at Institut de Cancérologie de l'Ouest well be included in this study.

Patients will be recruited in consultation before the start of reconstruction and up to 18 months after radiation therapy.

They will be followed for 24 months from the end of the breast reconstruction.

The following data will be collected indirectly from the clinical medical record (letters, reports of examinations, consultations, surgical report, hospitalization) of the patient, supplemented if necessary by specific records (radiotherapy records, chemotherapy, physiotherapy management) :

* Clinical data
* Technique-related data
* Complication-related data : adverse events will be evaluated at 15 days, 3 months, 6 months, 12 months and 24 months after reconstruction
* Aesthetic results data : aesthetic result will be evaluated by patients and surgeons at 6 months, 12 months and 24 months after reconstruction
* Quality of life data : a questionnaire will be submitted prior to the intervention, at 12 months and 24 months after reconstruction

Clinicians at Institut de Cancérologie de l'Ouest may be asked to complete the previous informations.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged over 18
* Medical history of mastectomy +/- radiotherapy
* Woman requesting breast reconstruction by implant
* Patient treated for non-metastatic cancer

Exclusion Criteria:

* Locally uncontrolled disease
* Metastatic disease
* Patient with major cutaneous atrophy allowing only flap reconstruction
* Patients under guardianship or trusteeship
* Patients who objected to the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns women who have had a mastectomy and want a secondary breast reconstruction by implant.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Describe the complications that occurs after a prepectoral placed implant with lipo-preparation | 12 months
  Pre-surgical implant positioning failure at 12 months. A failure will be defined by the occurence of at least one of the following complications : documented infection ; red breast syndrome ; hematoma ; lymphocele ; delayed healing ; prothesis removal ; stage 1 hull (Baker classification) ; prothesis rotation ; waves / folds ; muscle contractions with prothesis animation ; pain (EVA 4 or 5)

SECONDARY OUTCOMES:
Evaluate the aesthetic result | 6 months, 12 months and 24 months
  Aesthetic result will be assessed by giving a mark from 0 to 5 for the following categories : general breast appearance ; breast curve ; breast consistency ; breast volume Both clinician and patient will complete the evaluation.
Evaluate the quality of life | 24 months
  Patient satisfaction and quality of life will be assessed from Breast Q. The evaluation criteria will be the Breast Q score 24 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Victoire BRILLAUD-MEFLAH, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest René Gauducheau, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No